CLINICAL TRIAL: NCT00767897
Title: The Impact of the Human Papilloma Virus in Pediatric Chronic Kidney Disease, Dialysis, and Transplant Patients
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Corina Nailescu, Associate Professor of Clinical Pediatrics, Indiana University
Other Study IDs: 0807-02
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease; Dialysis
Keywords: Dose response relationship; immunity
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- CKD stage 3 or 4: Girls and Boys age 9-18 with CKD stage 3 or 4
  Interventions: Drug: Human Papillomavirus Vaccine
- On dialysis: Girls and Boys age 9-18 who are on dialysis
  Interventions: Drug: Human Papillomavirus Vaccine
- Transplanted: Girls and Boys age 9-18 who have had a functioning kidney transplant for longer than 6 months and are on the same immunosuppression regimen.
  Interventions: Drug: Human Papillomavirus Vaccine
- Healthy: Girls and Boys age 9-18
  Interventions: Drug: Human Papillomavirus Vaccine

INTERVENTIONS:
Drug: Human Papillomavirus Vaccine — The HPV vaccination will be administered by intramuscular injection in three separate 0.5mL doses. The recommended schedule is a 3-dose series with dose #2 and #3 administered 2 and 6 months after dose #1, respectively. The minimum interval between dose #1 and #2 of the vaccine is 4 weeks. The minimum recommended interval between dose #2 and #3 of the vaccine is 12 weeks.

SUMMARY:
The proposed study is a pilot study and a first step towards developing an optimized HPV vaccination strategy for girls who have CKD, or are on dialysis or have a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* 9-18-year-old girls who have CKD stages 3 or 4 (Glomerular filtration rates 15-59 mL/min/1.73m2).
* 9-18-year-old girls who are on dialysis.
* 9-18-year-old girls who have had a functioning kidney transplant for longer than 6 months and are on the same immunosuppression regimen.
* Healthy 9-18-year-old girls

Exclusion Criteria:

* Pregnancy, fever, allergy to any vaccine component, any immune disorder and any blood product received in the previous 6 months.

Ages: 9 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Girls age 9-18 who are healthy, have chronic kidney disease stage 3 or 4, are on dialysis, or have had a functioning kidney transplant for longer than 6 months and are on the same immunosuppression regimen.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corina Nailescu, M.D., Principal Investigator — Indiana University/Riley Children's Hospital
Locations (1):
- Indiana University/Riley Children's Hospital, Indianapolis, Indiana, United States